CLINICAL TRIAL: NCT03106363
Title: Effects of Combined Alcohol and Cannabis on Young Drivers' Simulated Driving
Brief Title: Combined Alcohol and Cannabis Effects on Skills of Young Drivers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Canada (Other Government)
Responsible Party: Principal Investigator, Christine Wickens, Independent Scientist, Institute for Mental Health Policy Research, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 123-2015
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Psychomotor Impairment
MeSH Terms: conditions — Psychomotor Disorders | interventions — Dronabinol; nabiximols; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Alcohol/Placebo Cannabis (Active Comparator): Participant will drink an alcoholic beverage to obtain a target blood alcohol content of 0.08mg% and will smoke a placebo delta 9 tetrahydrocannabinol (< 0.03%) cigarette.
  Interventions: Drug: placebo delta 9 tetrahydrocannabinol; Drug: Alcohol
- Placebo Alcohol/Cannabis (Active Comparator): Participant will drink tonic water (capped with a minimal amount of alcohol to enhance alcohol cues) and will smoke a delta 9 tetrahydrocannabinol (potency 12.5%) cigarette.
  Interventions: Drug: delta 9 tetrahydrocannabinol; Drug: Placebo alcohol
- Alcohol/Cannabis (Active Comparator): Participant will drink an alcoholic beverage to obtain a target blood alcohol content of 0.08mg% and will smoke a delta 9 tetrahydrocannabinol (potency 12.5%) cigarette.
  Interventions: Drug: delta 9 tetrahydrocannabinol; Drug: Alcohol
- Placebo Alcohol/Placebo Cannabis (Placebo Comparator): Participant will drink tonic water (capped with a minimal amount of alcohol to enhance alcohol cues) and will smoke a placebo delta 9 tetrahydrocannabinol (< 0.03%) cigarette.
  Interventions: Drug: placebo delta 9 tetrahydrocannabinol; Drug: Placebo alcohol

INTERVENTIONS:
Drug: delta 9 tetrahydrocannabinol — A single cannabis cigarette (potency 12.5% delta 9 tetrahydrocannabinol) will be given to participants to smoke over a 10 minute period, ad libitum. If the cannabis cigarette is not smoked in its entirety, the remainder will be weighed to estimate dose.
  Other Names: cannabis sativa; marijuana
  Arms: Alcohol/Cannabis; Placebo Alcohol/Cannabis
Drug: placebo delta 9 tetrahydrocannabinol — A single placebo cannabis cigarette (<0.03% delta 9 tetrahydrocannabinol) will be given to participants to smoke over a 10 minute period, ad libitum. If the placebo cannabis cigarette is not smoked in its entirety, the remainder will be weighed to estimate dose (as this is a double-blind study).
  Other Names: cannabis sativa; marijuana
  Arms: Alcohol/Placebo Cannabis; Placebo Alcohol/Placebo Cannabis
Drug: Alcohol — A single oral administration of an alcoholic beverage mixed in a 1:3 ratio of alcohol to tonic water to obtain a target blood alcohol content of 0.08mg%.
  Other Names: ethanol
  Arms: Alcohol/Cannabis; Alcohol/Placebo Cannabis
Drug: Placebo alcohol — A single oral administration of a beverage containing tonic water of the same volume as the alcoholic beverage.
  Other Names: Tonic water
  Arms: Placebo Alcohol/Cannabis; Placebo Alcohol/Placebo Cannabis

SUMMARY:
Alcohol and cannabis are the two most widely used substances of abuse in the world and are the psychoactive substances most often found in seriously and fatally injured drivers. In a recent study, it was observed that individuals who reported both driving under the influence of alcohol (DUIA) and the influence of cannabis (DUIC) experienced collision risk that was nearly 4 times that of individuals who reported driving after using only one of these drugs. Recent research in the United States and Canada indicates that the prevalence of DUIC among young drivers of high school and university age, and young adults is similar to, or higher than, the prevalence of DUIA. This is a serious public health issue, since motor vehicle collisions are the leading cause of death in this age group. Given the frequency with which alcohol and cannabis are consumed together, it is important to understand their combined effects on driver behaviour. The current study will examine the acute effects of a moderate dose of cannabis (12.5% THC) combined with an intoxicating amount of alcohol (BAC=0.08) on driving simulator performance of young drivers. Following an eligibility screening and practice session, a total of 70 participants aged 19 to 29 years will each complete 4 experimental sessions. During each session, participants will drink alcohol or placebo alcohol and smoke an active or placebo cannabis cigarette. The effects of alcohol and cannabis on the performance of driving-related skills will be assessed using a high-fidelity driving simulator. Cognitive, psychomotor, and mood effects will also be assessed.

DETAILED DESCRIPTION:
The proposed study will pursue the following primary aims:

Aim 1: Examine the acute effects of a moderate dose of cannabis (12.5% THC) combined with an intoxicating amount of alcohol (BAC=0.08) on driving simulator performance of young drivers. Simulated driving performance, tests of cognition, verbal memory, and mood will be measured concurrently with BAC and levels of cannabinoids in biological fluids before and after acute drug exposure in male and female drivers aged 19 to 29. BAC and biological fluids will be measured up to 5 hours following drug exposure.

Aim 2: Explore the effects of driving history, driving attitudes, and individual difference measures (e.g., demographics, drug and alcohol use, etc.) on the acute effects of alcohol and cannabis on driving simulator performance of young drivers. Exploratory analyses will be undertaken to determine if the acute effects of cannabis plus alcohol on the driving simulator task are influenced by these measures.

Study Design and Duration

This study will be a within-subjects, double-blind, double-dummy, placebo-controlled, counterbalanced, randomized clinical trial assessing the impact of alcohol and cannabis combined on driver behaviour. Although a placebo condition is part of the study, this is not a treatment study.

Initial contact with potential participants will be made via telephone, and study personnel will conduct a telephone screen for eligibility. Upon eligibility confirmation by telephone, participants will be asked to attend CAMH for an eligibility assessment. Participants will attend CAMH for a total of 6 study sessions (an eligibility assessment, a practice day, and 4 test sessions).

At each of four test sessions, participants will undergo one of these alcohol and cannabis exposure conditions: 1) placebo alcohol and placebo cannabis; 2) intoxicating dose of alcohol and placebo cannabis; 3) placebo alcohol and active cannabis, and; 4) intoxicating dose of alcohol and active cannabis. The order of these conditions will be randomly assigned. Participants will complete the alcohol manipulation followed by the cannabis manipulation. The alcohol and cannabis exposure sessions will be separated by at least 72 hours.

Participants will be asked not to use cannabis for 72 hours and alcohol for 48 hours prior to attending CAMH.

In certain instances, the Qualified Investigator may ask a participant to return for re-screening, e.g. repeat of urine test or other assessments performed for eligibility assessment. Also, in case of unforeseen delays in scheduling study participation, the Qualified Investigator will determine if there is a need to ask a participant to repeat some assessments, e.g., physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Use of cannabis at least once a week confirmed by urine point-of-care testing;
* Males who report consuming at least 5 drinks and females who report consuming at least 4 drinks in about 2 hours in the past 6 months and at least one episode of rapid alcohol consumption in the past 6 months (3 or more drinks over a span of one hour)
* 19-29 years of age;
* Holds a class G or G2 Ontario driver's licence (or equivalent from another jurisdiction) for at least 12 months;
* Willing to abstain from using alcohol for 48 hours and cannabis for 72 hours prior to Practice and Test Sessions.
* Willing to abstain from all other drugs not prescribed for medical purposes for the duration of the study;
* Provides written and informed consent.

Exclusion Criteria:

* Urine toxicology screens negative for cannabis upon eligibility assessment;
* Diagnosis of severe medical or psychiatric conditions;
* Females: Pregnancy or breastfeeding;
* Meets criteria for Alcohol or Substance Dependence (current or lifetime) (DSM-IV);
* Is a regular user of medications that affect brain function (i.e., antidepressants, benzodiazepines, stimulants);
* Taking medications or have any medical condition for which alcohol is contraindicated;
* First-degree relative diagnosed with schizophrenia;
* Severe allergy to citrus (lemon-lime).

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Psychomotor impairment: Standard deviation of lateral position | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Driving simulation tests occur within 2 hours before and approximately 45 minutes after Time 0.
  The driving simulator will objectively measure changes in driving behavior after alcohol and/or cannabis exposure.

SECONDARY OUTCOMES:
Psychomotor impairment: Mean speed, standard deviation of speed, and maximum speed | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Driving simulation tests occur within 2 hours before and approximately 45 minutes after Time 0.
  The driving simulator will objectively measure changes in driving behavior after alcohol and/or cannabis exposure.
Psychomotor impairment: Minimum time to collision and brake latency | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Driving simulation tests occur within 2 hours before and approximately 45 minutes after Time 0.
  The driving simulator will objectively measure changes in driving behavior after alcohol and/or cannabis exposure.
Psychomotor impairment: Number of collisions | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Driving simulation tests occur within 2 hours before and approximately 45 minutes after Time 0.
  The driving simulator will objectively measure changes in driving behavior after alcohol and/or cannabis exposure.
Subjective alcohol and cannabis effects | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Visual analogue scales are administered within 2 hours before as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Visual analogue scale measures how participants feel before and after alcohol and/or cannabis exposure.
Cognitive testing | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Cognitive testing is administered within 2 hours before Time 0 as well as approximately 75 minutes after Time 0.
  Measures changes in performance related to attention, memory, field of view, and dexterity before and after alcohol and/or cannabis exposure.
Breath alcohol content | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Breath alcohol content is measured within 2 hours before Time 0 as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Changes in BAC after drinking alcohol.
Blood concentration for delta 9 tetrahydrocannabinol, carboxy-tetrahydrocannabinol, and 11 hydroxy tetrahydrocannabinol. | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Blood concentration for THC, THC-COOH, and 11-OH-THC is assessed within 2 hours before Time 0 as well approximately 45 minutes after Time 0.
  Changes in concentration of delta 9 tetrahydrocannabinol (THC) , carboxy-tetrahydrocannabinol (THC-COOH), and 11 hydroxy tetrahydrocannabinol (11-OH-THC) in blood.
Urine cannabinoids corrected for creatinine | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Ratio of excreted THC metabolite carboxy-THC to creatinine is assessed within 2 hours before Time 0 as well as approximately 5 hours after Time 0.
  Determination of the ratio of excreted THC metabolite carboxy-THC to creatinine will determine whether participants have used cannabis between testing days, and hence will be excluded from further participation.
Vital signs: blood pressure | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Vital signs are assessed within 2 hours before as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Changes in blood pressure (systolic/diastolic)
Vital signs: pulse | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Vital signs are assessed within 2 hours before as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Changes in pulse
Vital signs: temperature | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Vital signs are assessed within 2 hours before as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Changes in temperature
Vital signs: respiration | Alcohol exposure is Time 0. Cannabis exposure follows 15 minutes after Time 0. Vital signs are assessed within 2 hours before as well as approximately 15, 30, 45, and 75 minutes and 2, 3, 4, and 5 hours after Time 0.
  Changes in respiration

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Wickens, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lenne MG, Dietze PM, Triggs TJ, Walmsley S, Murphy B, Redman JR. The effects of cannabis and alcohol on simulated arterial driving: Influences of driving experience and task demand. Accid Anal Prev. 2010 May;42(3):859-66. doi: 10.1016/j.aap.2009.04.021. PMID 20380913
- [Background] Downey LA, King R, Papafotiou K, Swann P, Ogden E, Boorman M, Stough C. The effects of cannabis and alcohol on simulated driving: Influences of dose and experience. Accid Anal Prev. 2013 Jan;50:879-86. doi: 10.1016/j.aap.2012.07.016. Epub 2012 Aug 4. PMID 22871272
- [Derived] Di Ciano P, Brands B, Fares A, Wright M, Stoduto G, Byrne P, McGrath M, Hasan OSM, Le Foll B, Wickens CM. The Utility of THC Cutoff Levels in Blood and Saliva for Detection of Impaired Driving. Cannabis Cannabinoid Res. 2023 Jun;8(3):408-413. doi: 10.1089/can.2022.0187. Epub 2023 Feb 2. PMID 36730769
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research